CLINICAL TRIAL: NCT02783183
Title: A Open-label, Radomized, Crossover Clinical Trial to Assess the Pharmacokinetics of Pregabalin CR After Multiple Dosing as Compared to Pregabalin IR in Healthy Male Volunteers
Brief Title: A Open-label, Randomized, Crossover Study to Assess PK of Pregabalin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: YHD1119-103
Record Dates: First submitted 2016-05-23; First posted 2016-05-26 (Estimated); Last update posted 2019-01-16 (Actual); Status verified 2016-11

CONDITIONS: Peripheral Nueropathy Pain
MeSH Terms: interventions — Pregabalin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- YHD1119 (Experimental): Pregabalin 300mg
  Interventions: Drug: YHD1119; Drug: Lyrica
- Lyrica (Active Comparator): Pregabalin 150mg
  Interventions: Drug: YHD1119; Drug: Lyrica

INTERVENTIONS:
Drug: YHD1119 — 2 by 2
  Other Names: Pregabalin 300mg
Drug: Lyrica — 2 by 2
  Other Names: Pregabalin 150mg

SUMMARY:
The purpose of this trial to compare the pharmacokinetic characteristics of YHD1119(Pregabalin 300mg) and Lyrica capsule(Pregabalin 150mg). YHD1119 is controlled release formulation which is made by Yuhan Corporation. Primary endpoints are Cmax,ss and AUCtau and secondary endpoints are AUClast,ss, AUCinf,ss, Tmax,ss and t1/2.

ELIGIBILITY:
Inclusion Criteria:

* 19~50 years old, healthy male volunteers
* >55Kg(Body weight) and 18.5<BMI<28

Exclusion Criteria:

* AST or ALT > 3 * Upper normal range (Lab)
* Total bilirubin > 2.0 mg/dl
* Systolic BP >140 OR <90, Diastolic BP >100 OR <60

Ages: 19 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2016-06; Primary Completion 2016-08 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Cmax,ss | 0.33,0.67,1,2,4,8,12,12.33,12.67,13,14,16,20,24,36 hours
AUCtau | 0.33,0.67,1,2,4,8,12,12.33,12.67,13,14,16,20,24,36 hours

SECONDARY OUTCOMES:
AUClast,ss | 0.33,0.67,1,2,4,8,12,12.33,12.67,13,14,16,20,24,36 hours
AUCinf,ss | 0.33,0.67,1,2,4,8,12,12.33,12.67,13,14,16,20,24,36 hours
Tmax,ss | 0.33,0.67,1,2,4,8,12,12.33,12.67,13,14,16,20,24,36 hours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Moon SJ, Jeon JY, Lim Y, An T, Jang SB, Kim S, Na WS, Lee SY, Kim MG. Pharmacokinetics of a New, Once-Daily, Sustained-release Pregabalin Tablet in Healthy Male Volunteers. Clin Ther. 2021 Aug;43(8):1381-1391.e1. doi: 10.1016/j.clinthera.2021.06.010. Epub 2021 Jul 11. PMID 34256964